CLINICAL TRIAL: NCT06950294
Title: High Dose Inhaled Nitric Oxide Therapy in Critically Ill Patients With Pneumonia: a Pilot, Double-blinded, Randomized, Controlled Trial
Brief Title: iNO300 Therapy in Critically Ill Patients With Pneumonia
Acronym: iNO300
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Lorenzo Berra, MD, Clinician Investigator, Associate Professor, Anesthesia, Critical Care and Pain Medicine, Mass General Research Institute, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2025P000909
Record Dates: First submitted 2025-04-13; First posted 2025-04-30 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Critical Illness; Pneumonia
Keywords: High dose inhaled nitric oxide; Pneumonia; Critical care; Methemoglobin
MeSH Terms: conditions — Critical Illness; Pneumonia | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- iNO300 group (Experimental): High dose inhaled nitric oxide starting at 250 ppm (not exceeding 300 ppm) , 40min, 4 times daily, from day 1 to day 5. Nitric oxide is delivered using a gas cylinder containing nitric oxide and nitrogen.
  Interventions: Drug: High dose inhaled nitric oxide; Other: standard therapy
- Control group (Sham Comparator): Sham intervention with the nitric oxide gas cylinder replaced by that containing only nitrogen and all other delivery procedures identical to the intervention group
  Interventions: Other: Sham treatment; Other: standard therapy

INTERVENTIONS:
Drug: High dose inhaled nitric oxide — Inhaled nitric oxide starting at 250-300 ppm, 40min, every 6 hours, from day 1 to day 5. Nitric oxide is delivered using a gas cylinder containing nitric oxide and nitrogen.
  Arms: iNO300 group
Other: Sham treatment — Sham intervention with the nitric oxide gas cylinder replaced by that containing only nitrogen and all other delivery procedures identical to the intervention group
  Arms: Control group
Other: standard therapy — Standard therapy pneumonia and critical illness

SUMMARY:
The goal of this clinical trial is to learn the formation and recovery rate of methemoglobin (MetHb) in severely sick patients with pneumonia who receive high doses of inhaled nitric oxide (iNO) therapy at 250 parts per million (ppm), not exceeding 300 ppm. Meanwhile, the benefits of the therapy to treat severely sick patients with pneumonia will be explored. Patients who are 18 years or older, newly diagnosed with pneumonia, and severely sick with requirement of a breathing machine could be included. The main questions it aims to answer are:

How does methemoglobin change through the iNO treatment? Does iNO therapy increase the number of patients recovering from pneumonia? Researchers will compare iNO treatment to placebo, which means using the same device as the treatment group without delivering the study drug.

Participants will:

* Receive iNO treatment starting at 250 ppm, not exceeding 300 ppm, 40 min, every 6 hours, from day 1 to day 5
* Be followed up for 60 days

DETAILED DESCRIPTION:
This study is designed as a pilot, double-blinded, randomized controlled trial to investigate levels of methemoglobin in the treatment group versus the control group and efficacy of high dose inhaled NO among critically ill patients with pneumonia. We will enroll 34 adult patients with newly diagnosed pneumonia and invasive mechanical ventilation who are admitted to the ICUs at Massachusetts General Hospital.

After enrollment, participants will be randomized in 1:1 ratio to intervention group or control group. Baseline characteristics will be collected.

During treatment period, patients allocated to the intervention group will receive high dose inhaled NO starting at 250 ppm (not exceeding 300 ppm), 40min, 4 times daily, for 5 days. The control group will receive sham intervention. Both groups will receive standard therapy.

During follow-up period, we will follow participants for a total duration of 60 days. Methemoglobin kinetic levels and efficacy outcomes will be collected.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Intubated and mechanically ventilated
* Within 72h of diagnosis of community- or hospital-acquired pneumonia
* Written informed consent obtained from patients or legally authorized representatives

Exclusion Criteria:

* Baseline methemoglobin 3% or higher
* Genetic diseases including glucose-6-phosphate dehydrogenase deficiency, cytochrome b5 reductase deficiency, sickle cell disease
* Oxygen saturation < 88% on 100% inspired fraction of oxygen
* Anemia with hemoglobin < 7.0 g/dl
* Acute cardiogenic shock requiring inotropic or mechanical support with an ejection fraction less than 20%
* eGFR < 30 ml/min/1.73m2 or use of continuous renal replacement therapy
* Receiving inhaled NO therapy or decision to initiate inhaled NO therapy within 24 hours post randomization
* A decision to do-not-resuscitate (DNR)
* Enrollment in another experimental antimicrobial treatment protocol
* Patients for whom follow-up is expected to be impossible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Peaks of methomoglobin | From Day 1 to Day 5
  Continuous recording of MetHb and peaks of MetHb will be determined.

SECONDARY OUTCOMES:
Nitrogen dioxide level | From Day 1 to Day 5
  Continuous measurement of nitrogen dioxide concentration in the inspiratory limb of breathing circuit
Feasibility | From enrollment to Day 60
  Referral, recruitment, retention, compliance and follow-up completion rates of the study
Clinical cure rate of pneumonia | From enrollment to test of cure day (4 -11 days post end of treatment)
  Clinical cure is assessed at test of cure (4 -11 days post end of treatment) and defined as resolution of clinical signs and symptoms of pneumonia compared with baseline, including a reduction in SOFA and CPIS scores, improvement or lack of progression in chest imaging, and no requirement for additional antibacterial treatment.
Clinical improvement rate of pneumonia | Day 5
  Clinical improvement is assessed at end of treatment and defined as improvement in 2 or more clinical signs and symptoms of pneumonia compared with baseline, improvement or lack of progression of chest x-ray abnormalities, and no requirement for additional antibacterial treatment. Clinical signs and symptoms of pneumonia include new onset or worsening cough, purulent sputum or increased suction requirements, auscultation findings of pneumonia, dyspnea, tachypnea, or respiratory rate ≥ 30/min, hypoxemia, worsening gas exchange.
Microbiologic eradication rate | From enrollment to test of cure day (4 -11 days post end of treatment)
  Absence of the baseline pathogen from tracheal aspiration or bronchoalveolar lavage fluid will be confirmed. If it is not possible to obtain an appropriate clinical specimen for culture and the patient has a successful clinical outcome, the response was presumed to be eradication.
28-day all cause mortality | From enrollment to Day 28
  All cause mortality from enrollment to Day 28
60-day all cause mortality | From enrollment to Day 60
  All cause mortality from enrollment to Day 60
28-day ventilator free days | From enrollment to Day 28
  Successful liberation from mechanical ventilation should last more than 48 h without re-intubation in patients who have survived 28 days after randomization (extubation was counted from the last successful attempt in patients who have survived 28 days since randomization) and for patients ventilated for 28 days or more or who died before 28 days (irrespective of intubation status), the number of ventilator-free days was recorded at zero.
Days free from organ support in 28 days | From enrollment to Day 28
  Organ support includes mechanical ventilation, vasopressors and renal replacement therapy.
Blood stream infection | From enrollment to Day 28
  Positive blood culture with a pathogenic bacterium
Days free from antibiotics during hospitalization | From enrollment to the day of hospital discharge or death, whichever comes earlier, assessed up to 60 days
  Days free from antibiotics during hospitalization
Acquisition of multidrug-resistant (MDR) infection or colonization | From enrollment to Day 28
  Multidrug-resistant infection is defined as pathogen acquiring non-susceptibility to at least one agent in three or more antibiotic categories
Hospital stay | From enrollment to the day of hospital discharge or death, whichever comes earlier, assessed up to 60 days
  Days from enrollment to the end of hospitalization
ICU length of stay | From enrollment to the day of ICU discharge or death, whichever comes earlier, assessed up to 60 days
  ICU length of stay
Inflammatory markers | From enrollment to test of cure (4-11 days post end of treatment)
  The test includes C reactive protein (CRP), procalcitonin (PCT), monocyte chemoattractant protein-1 (MCP-1), tumor necrosis factor α (TNF α), interleukin 6 (IL-6), interleukin 8 (IL-8), interleukin 10 (IL-10).

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Berra, MD, Principal Investigator — Anesthesia, Critical Care and Pain Medicine, Massachusetts General Hospital

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Beginning 1 year after publication with no end date
Access Criteria: A proposal that describes planned analyses must be submitted to the principal investigator via email. Data sharing agreement should be reached, documented and signed.

REFERENCES:
- [Background] Tal A, Greenberg D, Av-Gay Y, Golan-Tripto I, Feinstein Y, Ben-Shimol S, Dagan R, Goldbart AD. Nitric oxide inhalations in bronchiolitis: A pilot, randomized, double-blinded, controlled trial. Pediatr Pulmonol. 2018 Jan;53(1):95-102. doi: 10.1002/ppul.23905. Epub 2017 Nov 27. PMID 29178284
- [Background] Wolak T, Dicker D, Shifer Y, Grossman A, Rokach A, Shitrit M, Tal A. A safety evaluation of intermittent high-dose inhaled nitric oxide in viral pneumonia due to COVID-19: a randomised clinical study. Sci Rep. 2024 Jul 26;14(1):17201. doi: 10.1038/s41598-024-68055-w. PMID 39060420
- [Background] Miller C, Miller M, McMullin B, Regev G, Serghides L, Kain K, Road J, Av-Gay Y. A phase I clinical study of inhaled nitric oxide in healthy adults. J Cyst Fibros. 2012 Jul;11(4):324-31. doi: 10.1016/j.jcf.2012.01.003. Epub 2012 Apr 18. PMID 22520076
- [Background] Wiegand SB, Safaee Fakhr B, Carroll RW, Zapol WM, Kacmarek RM, Berra L. Rescue Treatment With High-Dose Gaseous Nitric Oxide in Spontaneously Breathing Patients With Severe Coronavirus Disease 2019. Crit Care Explor. 2020 Nov 16;2(11):e0277. doi: 10.1097/CCE.0000000000000277. eCollection 2020 Nov. PMID 33225304
- [Background] Strickland B, Albala L, Coffey EC, Carroll RW, Zapol WM, Ichinose F, Berra L, Harris NS. Safety and practicality of high dose inhaled nitric oxide in emergency department COVID-19 patients. Am J Emerg Med. 2022 Aug;58:5-8. doi: 10.1016/j.ajem.2022.04.052. Epub 2022 May 4. PMID 35623183
- [Background] Safaee Fakhr B, Di Fenza R, Gianni S, Wiegand SB, Miyazaki Y, Araujo Morais CC, Gibson LE, Chang MG, Mueller AL, Rodriguez-Lopez JM, Ackman JB, Arora P, Scott LK, Bloch DB, Zapol WM, Carroll RW, Ichinose F, Berra L; Nitric Oxide Study Investigators. Inhaled high dose nitric oxide is a safe and effective respiratory treatment in spontaneous breathing hospitalized patients with COVID-19 pneumonia. Nitric Oxide. 2021 Nov 1;116:7-13. doi: 10.1016/j.niox.2021.08.003. Epub 2021 Aug 13. PMID 34400339
- [Background] Wiegand SB, Traeger L, Nguyen HK, Rouillard KR, Fischbach A, Zadek F, Ichinose F, Schoenfisch MH, Carroll RW, Bloch DB, Zapol WM. Antimicrobial effects of nitric oxide in murine models of Klebsiella pneumonia. Redox Biol. 2021 Feb;39:101826. doi: 10.1016/j.redox.2020.101826. Epub 2020 Dec 11. PMID 33352464
- [Background] Valsecchi C, Winterton D, Safaee Fakhr B, Collier AY, Nozari A, Ortoleva J, Mukerji S, Gibson LE, Carroll RW, Shaefi S, Pinciroli R, La Vita C, Ackman JB, Hohmann E, Arora P, Barth WH Jr, Kaimal A, Ichinose F, Berra L; DELiverly oF iNO (DELFiNO) Network Collaborators. High-Dose Inhaled Nitric Oxide for the Treatment of Spontaneously Breathing Pregnant Patients With Severe Coronavirus Disease 2019 (COVID-19) Pneumonia. Obstet Gynecol. 2022 Aug 1;140(2):195-203. doi: 10.1097/AOG.0000000000004847. Epub 2022 Jul 6. PMID 35852269
- [Background] Bartley BL, Gardner KJ, Spina S, Hurley BP, Campeau D, Berra L, Yonker LM, Carroll RW. High-Dose Inhaled Nitric Oxide as Adjunct Therapy in Cystic Fibrosis Targeting Burkholderia multivorans. Case Rep Pediatr. 2020 Jun 24;2020:1536714. doi: 10.1155/2020/1536714. eCollection 2020. PMID 32685229
- [Background] Okda M, Spina S, Safaee Fakhr B, Carroll RW. The antimicrobial effects of nitric oxide: A narrative review. Nitric Oxide. 2025 Apr;155:20-40. doi: 10.1016/j.niox.2025.01.001. Epub 2025 Jan 8. PMID 39793728